CLINICAL TRIAL: NCT06534918
Title: Precise Oncology Interventions in Nutrition and Training (OnPoint)
Acronym: OnPoint
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: The Applebaum Foundation (Unknown)
Responsible Party: Principal Investigator, Tracy E Crane, PhD, RDN, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20230533
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Prostate Cancer; Colorectal Cancer
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Colorectal Neoplasms | interventions — Nutritional Status

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low Complexity Group (Experimental): Participants in this group will receive the low complexity intervention for up to eight (8) weeks.
  Interventions: Other: Fitbit; Behavioral: Nutrition and Physical Activity Prescription
- Moderate Complexity Group (Experimental): Participants in this group will receive the moderate complexity intervention for up to eight (8) weeks.
  Interventions: Other: Fitbit; Behavioral: Nutrition Course: Group Sessions; Behavioral: Physical Activity Program: Group Sessions; Behavioral: Nutrition and Physical Activity Prescription
- High Complexity Group (Experimental): Participants in this group will receive the high complexity intervention for up to eight (8) weeks.
  Interventions: Other: Fitbit; Behavioral: Nutrition Course: One on One Sessions with Registered Dietitian; Behavioral: Physical Activity Program: One on One Sessions with an Exercise Physiologist; Behavioral: Nutrition and Physical Activity Prescription
- Control Group (No Intervention): Participants randomized to this arm will receive routine care and will not receive any study materials until the end of the study at 24 weeks.

INTERVENTIONS:
Other: Fitbit — Participants will be provided with a Fitbit. Self-reported physical activity, location, vital sign and sleep stage information will be collected and monitored every day for up to eight (8) weeks. Data will be synced to the My Wellness Research Software Platform, resulting in a weekly text or phone call check-in, based on participants preference.
  Arms: High Complexity Group; Low Complexity Group; Moderate Complexity Group
Behavioral: Nutrition Course: Group Sessions — The nutrition course will follow a combined asynchronous and synchronous approach. The asynchronous component will consist of a pre-recorded session covering educational nutrition content, which will be made available to participants for self-paced learning. This will be followed by a synchronous, 30-60 minute live group education class on nutrition information for cancer survivors, held once per week.
  Arms: Moderate Complexity Group
Behavioral: Physical Activity Program: Group Sessions — The Physical Activity Program will be held virtually or in-person. This will be a 1-hour biweekly group education class on aerobic and resistance exercise recommendations for cancer survivors.
  Arms: Moderate Complexity Group
Behavioral: Nutrition Course: One on One Sessions with Registered Dietitian — Participants will be referred to weekly one on one nutrition counseling sessions with a Registered Dietitian. The one on one sessions are anticipated to last 30-60 minutes, based on the needs of the individual.
  Arms: High Complexity Group
Behavioral: Physical Activity Program: One on One Sessions with an Exercise Physiologist — Participants will be referred to weekly one on one exercise training sessions with an Exercise Physiologist. The one on one sessions are anticipated to last 30-60 minutes, based on the needs of the individual
  Arms: High Complexity Group
Behavioral: Nutrition and Physical Activity Prescription — Participants will receive a lifestyle medicine prescription pad, developed by the investigators, which serves as a checklist to assist participants in effectively monitoring their dietary habits and physical activity routines. Participants will also receive an 8-week text messages program which will direct participants to a webpage with nutrition and physical activity content.
  Arms: High Complexity Group; Low Complexity Group; Moderate Complexity Group

SUMMARY:
The purpose of this study is to see if survivors of breast, prostate, or colorectal cancer who receive a personal referral to a targeted nutrition and exercise program will be able to eat a healthier diet and be more physically activity.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria - Healthcare Providers

1. Provide full- or part-time care in an oncology clinical care setting at Sylvester Comprehensive Cancer Center
2. Utilize the electronic medical record for patient documentation on a regular basis
3. Willing to complete a 30-60-minute interview

Inclusion Criteria - Patients

1. 18 years of age or older
2. Any sex/gender
3. Able to provide consent
4. Able to read/understand English or Spanish
5. Diagnosis of breast, prostate or colorectal cancer, 6 months post completion of primary treatment, with no evidence of primary disease
6. Approval from treating oncologist, confirmed via email or in writing
7. Fail to meet at least one of the American Cancer Society guidelines: engaging in >150 minutes of moderate-to-vigorous physical activity per week for the prior month or consuming at least 3 cups of vegetables and 2 cups of fruit per day over the past month.
8. Internet access on a smart phone, tablet, or computer
9. Agree to be randomly assigned to any study group

Exclusion Criteria:

1. Less than 18 years of age
2. Unable to provide consent
3. Unable to read/understand English or Spanish
4. Any contraindication for diet change or exercising as determined by physician
5. Blank
6. Engaging in >150 minutes of moderate to vigorous physical activity on average per week for the prior month
7. Meeting the American Cancer Society diet recommendations (3 cups of vegetables or legumes, 2 cups of fruit, 2 serving whole grain per day, and limited red/processed meats, sugar-sweetened beverages, and highly processed foods) for the prior month
8. History of dementia or major psychiatric disease which would interfere with study participation
9. History of recent (≤1 yr) stroke, myocardial infarction or congestive heart failure
10. Eastern Cooperative Oncology Group (ECOG) score of >2
11. Severe lymphedema as determined by physician
12. Receiving physical therapy treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Survivors Who Agree to Participate | Up to 8 Weeks
  Percentage of survivors who agree to participate will be reported as ≥ 50%.
Percentage of Interventions Sessions Completed | Up to 8 Weeks
  Percentage of intervention sessions completed will be reported as ≥ 80%.
Percentage of Participants Satisfied with the Intervention | Up to 8 Weeks
  Report of 80% satisfaction will be determined as satisfaction with intervention components.

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Crane, PhD, RDN, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No